CLINICAL TRIAL: NCT01623401
Title: Phase 1, Open-Label, Ophthalmology and Neurology Safety Study of Oral 200 mg TR-701 FA Once Daily for 10 Days in Healthy Adults
Brief Title: A Phase 1, Open-Label, 10 Day Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1986-030; TR701-110 (Other: TriusRX unique ID)
Record Dates: First submitted 2012-06-06; First posted 2012-06-20 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — tedizolid phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TR-701 FA (Experimental): TR-701 FA 200 mg oral once daily
  Interventions: Drug: TR-701 FA

INTERVENTIONS:
Drug: TR-701 FA — TR-701 FA 200 mg once daily
  Other Names: Tedizolid Phosphate

SUMMARY:
This is a Phase 1 open-label study in healthy volunteers who will receive oral 200 mg TR 701 FA once daily for 10 days and will include ophthalmologic and neurologic assessments.

DETAILED DESCRIPTION:
This is a Phase 1 open-label study in healthy volunteers who will receive oral 200 mg TR 701 FA once daily for 10 days (Days 1 through 10) and undergo safety evaluations including ophthalmologic and neurologic assessments before (Screening or Day -1), 1 day after final study drug administration (Day 11 or earlier if a subject discontinues treatment), and 2 to 4 weeks after the last study drug administration (Late Follow-up Visit).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females ≥ 18 and ≤ 65 years of age with no clinically significant abnormalities identified by a detailed medical history
* Female subjects must be nonpregnant, nonlactating, and either postmenopausal for at least 2 years, surgically sterile for at least 90 days, abstinent, or agree to use contraception from 1 week prior to Day -1 until 30 days after leaving the study center.
* Male subjects must be surgically sterile, abstinent, or agree to use contraception from Day -1 until 30 days after leaving the study center
* BMI ≥ 18.0 kg/m2 and ≤ 35.0 kg/m2

Exclusion Criteria:

* Hypersensitivity to oxazolidinones or any component in the formulation
* History or current significant ophthalmologic or neurologic condition that would adversely affect the clinical assessments or confound the interpretation of the data (e.g., dense cataracts, macular degeneration, retinitis pigmentosa)
* Positive hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus antibody test result
* Known genetic condition related to mitochondrial disease or dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-05-17 (Actual); Primary Completion 2012-08-24 (Actual); Study Completion 2012-08-24 (Actual)

PRIMARY OUTCOMES:
Safety | 6 weeks
  The primary objective is to determine the safety of oral 200 mg TR-701 free acid (FA) administered once daily for 10 days in healthy adults. Safety outcome measures include the number and proportion of participants with adverse events, changes in vital signs and ECG, and evaluation of physical examination changes including neurologic and ophthalmologic exams.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (1):
- Trius Investigator Site 001, Dallas, Texas, United States

REFERENCES:
- [Result] Fang E, Munoz KA, Prokocimer P. Characterization of Neurologic and Ophthalmologic Safety of Oral Administration of Tedizolid for Up to 21 Days in Healthy Volunteers. Am J Ther. 2017 Mar/Apr;24(2):e227-e233. doi: 10.1097/MJT.0000000000000534. PMID 27941424